CLINICAL TRIAL: NCT01364441
Title: A Double-Blind, Placebo-Controlled, Single-Dose Escalation and Food Effect Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ONO-2952 in Healthy Adult Subjects
Brief Title: Single-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ONO-2952 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Organization: Ono Pharmaceutical Co. Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-2952POU001
Record Dates: First submitted 2011-05-25; First posted 2011-06-02 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Healthy Adult Subjects
Keywords: ONO-2950; healthy adult subjects; first in human; safety; tolerability; pharmacokinetics
MeSH Terms: interventions — ONO-2952

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- P (Placebo Comparator)
  Interventions: Drug: Placebo
- E (Experimental)
  Interventions: Drug: ONO-2952

INTERVENTIONS:
Drug: ONO-2952 — 3 mg to 800 mg at a single dose; 10 mg and 200 mg for food effect study
  Arms: E
Drug: Placebo — Placebo dosed in the same manner as ONO-2952
  Arms: P

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of ONO-2952 across ascending single doses in healthy adult male and female subjects. The secondary objective is to characterize the pharmacokinetic (PK) profile of ONO-2952. The tertiary objective of this study is to preliminarily evaluate the effect of a meal upon the PK profile of ONO-2952.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking male or female subjects (18-55 inclusive)
* Body mass index (BMI) of 19-35 kg/m2 (inclusive)
* For females, surgically sterilized, postmenopausal, or who are non- lactating and agree to use a double barrier method of contraception

Exclusion Criteria:

* History or presence of clinically significant disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ONO-2952 using vital signs, ECGs, laboratory tests, physical examinations, and incidence/severity of adverse events | up to 8 days

SECONDARY OUTCOMES:
Characterization of PK of ONO-2952 through measurement of drug concentration in plasma and urine sample | up to 8 days
Effect of food on ONO-2952 pharmacokinetics by comparison of PK profile between fasted and fed conditions | up to 24 days

CONTACTS AND LOCATIONS:
Overall Officials: Ono Pharma USA, Inc., Study Director — Ono Pharmaceutical Co. Ltd
Locations (1):
- Austin Clinical Site, Austin, Texas, United States

REFERENCES:
- [Derived] Suto F, Wood AT, Kobayashi M, Komaba J, Duffy K, Bruce M. Safety, Tolerability, and Pharmacokinetic Profile of the Novel Translocator Protein 18 kDa Antagonist ONO-2952 in Healthy Volunteers. Clin Ther. 2015 Sep;37(9):2071-84. doi: 10.1016/j.clinthera.2015.07.010. Epub 2015 Aug 4. PMID 26249232